CLINICAL TRIAL: NCT00245102
Title: A Multicenter Phase II Study of Sorafenib (BAY43-9006) in Non-GIST Sarcomas
Brief Title: Sorafenib in Treating Patients With Metastatic, Locally Advanced, or Recurrent Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01469; NCI-2012-01469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-7060; CDR0000449962; MSKCC-05081; 05-081 (Other: Memorial Sloan-Kettering Cancer Center); 7060 (Other: CTEP); N01CM62206 (NIH); P30CA008748 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2012-12

CONDITIONS: Adult Angiosarcoma; Adult Epithelioid Sarcoma; Adult Leiomyosarcoma; Adult Malignant Fibrous Histiocytoma; Adult Neurofibrosarcoma; Adult Synovial Sarcoma; Ovarian Sarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Uterine Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage III Uterine Sarcoma; Stage IV Adult Soft Tissue Sarcoma; Stage IV Uterine Sarcoma; Uterine Carcinosarcoma; Uterine Leiomyosarcoma
MeSH Terms: conditions — Hemangiosarcoma; Sarcoma; Leiomyosarcoma; Histiocytoma, Malignant Fibrous; Neurofibrosarcoma; Sarcoma, Synovial | interventions — Sorafenib

ARMS (1):
- Arm I (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with metastatic, locally advanced, or recurrent sarcoma. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary endpoint is the response rate (CR+PR) for each stratum of sarcoma patients treated with sorafenib as defined by RECIST.

SECONDARY OBJECTIVES:

I. Progression-free survival (defined as CR + PR + SD, assessed at 3 months or 6 months).

II. Overall survival. III. Pharmacokinetics of sorafenib in this patient population (all sites will participate).

IV. Frequency of B-raf mutations in the patients' sarcomas treated as part of this study and correlation with response or resistance to sorafenib (all sites will participate).

V. Ras-raf kinase pathway activation in pre-treatment existing tumor specimens (paraffin section immunohistochemistry; all sites will participate).

VI. At MSKCC only: Pre and post treatment specimen changes in downstream events of ras signaling, specifically inhibition of ERK phosphorylation. Only patients with angiosarcoma and MPNST will undergo biopsy (up to 10 patients).

VII. At MSKCC only: Circulating Endothelial Cells (CECs), VE-cadherin levels, and soluble protein levels (VEGF, bFGF, endostatin) as a measures of angiogenesis before and after starting sorafenib therapy.

OUTLINE: This is an open-label, non-randomized, multicenter study. Patients are stratified according to sarcoma histology (angiosarcoma vs malignant peripheral nerve sheath tumor vs leiomyosarcoma [closed to accrual as of 11/29/06] vs high-grade undifferentiated pleomorphic sarcoma [i.e., malignant fibrous histiocytoma (including myxofibrosarcoma)(closed to accrual as of 11/29/06)] vs synovial sarcoma (closed to accrual as of 11/29/06) vs all other types of sarcoma).

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed sarcoma, including any of the following neoplastic subtypes:

  * Giant hemangioma
  * Angiosarcoma (including epithelioid hemangioendothelioma)
  * Malignant peripheral nerve sheath tumor
  * Leiomyosarcoma (closed to accrual as of 11/29/06)
  * High-grade undifferentiated pleomorphic sarcoma (i.e., malignant fibrous histiocytoma [including myxofibrosarcoma]) (closed to accrual as of 11/29/06)
  * Synovial sarcoma (closed to accrual as of 11/29/06)
  * Carcinosarcoma (closed to accrual as of 11/29/06)
* Metastatic, locally advanced, or locally recurrent disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Lesions in a previously irradiated area may be considered measurable provided there is evidence of subsequent disease progression that cannot be attributed to necrosis or bleeding
* No gastrointestinal stromal tumor
* No known brain metastases
* Performance status - ECOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No evidence of bleeding diathesis
* Bilirubin ≤ 1.5 mg/dL
* INR ≤ 1.5
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension
* No history of allergic reaction to compounds of similar chemical or biologic composition to sorafenib
* No known HIV positivity
* No active or ongoing infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness or social situation that would preclude study compliance
* No swallowing dysfunction that would preclude the swallowing of tablets
* Other malignancies allowed provided sarcoma is the primary disease requiring treatment
* No other uncontrolled illness
* No more than 1 prior chemotherapy regimen for recurrent or metastatic disease (≤ 3 regimens for angiosarcoma or malignant peripheral nerve sheath tumor)

  * Adjuvant chemotherapy completed > 1 year prior to study entry is not considered a line of prior treatment
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* At least 3 weeks since prior radiotherapy
* Recovered from prior antitumor therapy

  * Alopecia allowed
* No prior sorafenib
* No prior small molecule inhibitors of MAPK signaling intermediates
* No concurrent therapeutic anticoagulation

  * Prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial devices allowed provided requirements for PT, INR, or PTT requirements are met
* No other concurrent investigational agents
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent rifampin or Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 09/09/2005 Protocol Closed to Accrual 07/22/2008 Primary Completion Date 03/22/2011 Recruitment Location is the medical clinic
Groups:
- Angiosarcoma; MPNST; Leiomyosarcoma; Undifferentiated Pleomorphic Sarcoma; Fibrosarcoma; Other Histology: Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Angiosarcoma | MPNST | Leiomyosarcoma | Undifferentiated Pleomorphic Sarcoma | Fibrosarcoma | Other Histology
Started | 44 | 16 | 46 | 13 | 5 | 23
Completed | 37 | 12 | 39 | 10 | 5 | 19
Not Completed | 7 | 4 | 7 | 3 | 0 | 4
Not completed — Not Treated | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 5 | 1 | 0 | 2
Not completed — Decline in performance | 0 | 2 | 0 | 1 | 0 | 2
Not completed — Participant needed surgery | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Clinical progression | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Angiosarcoma; MPNST; Leiomyosarcoma; Undifferentiated Pleomorphic Sarcoma; Fibrosarcoma; Other Histology: Sorafenib 400 mg PO BID
- Total: Total of all reporting groups
Arm/Group | Angiosarcoma | MPNST | Leiomyosarcoma | Undifferentiated Pleomorphic Sarcoma | Fibrosarcoma | Other Histology | Total
Number analyzed (Participants) | 44 | 16 | 46 | 13 | 5 | 23 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 14 | 35 | 7 | 5 | 22 | 103
  >=65 years | 24 | 2 | 11 | 6 | 0 | 1 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (50.91168825) | 47.5 (34.64823228) | 56 (33.9411255) | 62.5 (31.81980515) | 43.5 (10.60660172) | 44 (31.11269837) | 54 (50.91168825)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 9 | 37 | 8 | 4 | 11 | 94
  Male | 19 | 7 | 9 | 5 | 1 | 12 | 53
Region of Enrollment [Number; unit: participants]
  United States | 44 | 15 | 46 | 13 | 5 | 23 | 146
  Italy | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Measured by Complete Response (CR) Rate and Partial Response (PR) Rate as Determined by RECIST
Description: A 5% response rate is considered not promising, a 20% response rate is considered promising. For each stratum, the response rate will be estimated and a confidence interval will be constructed.
Time Frame: Up to 4 weeks
Measure: Number; unit: participants
Arm/Group | Angiosarcoma | MPNST | Leiomyosarcoma | Undifferentiated Pleomorphic Sarcoma | Fibrosarcoma | Other Histology
Number analyzed (Participants) | 37 | 12 | 39 | 10 | 5 | 19
participants
  Complete Response | 1 | 0 | 0 | 0 | 0 | 0
  Partial Response | 4 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Angiosarcoma | MPNST | Leiomyosarcoma | Undifferentiated Pleomorphic Sarcoma | Fibrosarcoma | Other Histology
Serious Adverse Events (participants affected / at risk) | 13/44 | 7/16 | 7/46 | 9/13 | 0/5 | 5/23
Other Adverse Events (participants affected / at risk) | 36/44 | 12/16 | 40/46 | 10/13 | 4/5 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Angiosarcoma (N=44) | MPNST (N=16) | Leiomyosarcoma (N=46) | Undifferentiated Pleomorphic Sarcoma (N=13) | Fibrosarcoma (N=5) | Other Histology (N=23)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death-Disease progression (General disorders) | 1/1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Anemia) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vision-flashing lights (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General symptom, other-Failure to thrive (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death, NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhage, Respiratory tract (NOS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hemorrhage, bleeding other-Chest wall (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiosarcoma (N=44) | MPNST (N=16) | Leiomyosarcoma (N=46) | Undifferentiated Pleomorphic Sarcoma (N=13) | Fibrosarcoma (N=5) | Other Histology (N=23)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Fatigue (General disorders) | 11 (11) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 7 (7) | 3 (3) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 3 (3) | 2 (24) | 3 (3) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 8 (8) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
INR increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 1 (1) | 6 (6) | 2 (2) | 1 (1) | 4 (4)
Lymphocyte count decreased (Investigations) | 7 (7) | 2 (2) | 7 (7) | 4 (4) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (12) | 1 (1) | 7 (7) | 2 (2) | 0 (0) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0) | 12 (12) | 2 (2) | 3 (3) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (15) | 5 (5) | 17 (17) | 2 (2) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary-Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decrease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less